CLINICAL TRIAL: NCT02823379
Title: Smart Walk: A Physical Activity Program for African American Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00003131; K99HL129012 (NIH); R00HL129012 (NIH)
Record Dates: First submitted 2016-07-01; First posted 2016-07-06 (Estimated); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Physical Activity
Keywords: physical activity; overweight; obese; exercise; women; African American; Smartphone; cardiovascular disease risk
MeSH Terms: conditions — Motor Activity; Overweight; Obesity | interventions — Exercise; Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical Activity (Experimental): A culturally relevant physical activity promotion program delivered using a Smartphone application.
  Interventions: Behavioral: Physical Activity
- Wellness Contact Control (Active Comparator): A wellness contract control condition delivered using a Smartphone application.
  Interventions: Behavioral: Wellness

INTERVENTIONS:
Behavioral: Physical Activity — A Smartphone delivered physical activity program
  Arms: Physical Activity
Behavioral: Wellness — A Smartphone delivered wellness intervention focused on topics other than physical activity (e.g., skin care, oral health, and breast exams).
  Arms: Wellness Contact Control

SUMMARY:
The purpose of this project is to test an 8-month, culturally relevant, Smartphone-delivered PA program to improve and maintain high physical levels and reduce cardiometabolic disease risk among obese AA women.

DETAILED DESCRIPTION:
A three-phase study will be used to refine and implement an established theory-based culturally relevant physical activity promotion intervention for obese African American women. Phase 1 (Aim 1a) will include formative research where 25 African American women provide feedback (via 9 focus groups) to further refine the physical activity intervention by specifying the deep structure cultural relevance of the theoretical mediators of self-regulation, self-efficacy, social support, behavioral capability, and outcome expectations.5 Phase 2 will focus on technical development of the refined culturally tailored intervention and 1-month demonstration trial of the Smartphone-delivered physical activity promotion program. Phase 3 (Aims 1b and 1c) will test the intervention and delivery strategy in a two-arm randomized trial where 60 sedentary, obese African American women will receive either the 8-month culturally relevant smartphone-delivered physical activity intervention or a 8-month wellness contact control condition

ELIGIBILITY:
Inclusion Criteria:

* Self-reported African American
* Insufficiently Active ( 60 mins or less of PA per wk measured by Exercise Vital Sign Questionnaire)
* BMI>30
* English speaking and reading
* Own non-Kindle Smartphone iOS 7 or above, or Android 2.3 or above

Exclusion Criteria:

* Concurrent participation in another physical activity, nutrition, or weight loss program
* Endorsement of an item on the Physical Activity Readiness Questionnaire (PAR-Q) unless physical note is provided
* Pregnant or plans to become pregnant in next 12 months
* Plans to relocate out of Phoenix area in next 12 months

Ages: 24 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2015-09; Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Change in physical activity from baseline to 8-months | three assessment periods: baseline, 4-months, and 8-months
  assessed by ActiGraph accelerometers
Feasibility and acceptability of the Smartphone delivered physical activity program | 4-months
  Feasibility and acceptability will be assessed by examining recruitment, retention, adherence, self-reported treatment acceptance, and participant utilization of the Smartphone application provided by analytic tracking software.

SECONDARY OUTCOMES:
change in body mass index (BMI) from baseline to 8-months | three assessment periods: baseline, 4-months, and 8-months
change in cardiorespiratory fitness from baseline to 8-months | three assessment periods: baseline, 4-months, and 8-months
  A modified Balke treadmill protocol will be used to estimate aerobic capacity (VO2peak).
change in Aortic Pulse Wave Velocity from baseline to 8-months | three assessment periods: baseline, 4-months, and 8-months
  A measure of aortic stiffness, will be assessed with SphymocorTM using validated methodology
change in blood pressure from baseline to 8-months | three assessment periods: baseline, 4-months, and 8-months
change in total serum cholesterol from baseline to 8-months | three assessment periods: baseline, 4-months, and 8-months
change in serum high-density lipoprotein (HDL) from baseline to 8-months | three assessment periods: baseline, 4-months, and 8-months
change in serum low-density lipoprotein (LDL) from baseline to 8-months | three assessment periods: baseline, 4-months, and 8-months
change in serum triglycerides from baseline to 8-months | three assessment periods: baseline, 4-months, and 8-months
change in serum insulin from baseline to 8-months | three assessment periods: baseline, 4-months, and 8-months
  measured using Immulite 1000 immunoassay analyzer (Siemens Healthcare Diagnostics)
change in insulin sensitivity from baseline to 8-months | three assessment periods: baseline, 4-months, and 8-months
  assessed by calculating homeostatic model assessment (HOMA) scores as: glucose (mg/dl) x insulin (μU/ml)/405.
change in tumor necrosis factor alpha from baseline to 8-months | three assessment periods: baseline, 4-months, and 8-months
change in Interleukin 1 beta from baseline to 8-months | three assessment periods: baseline, 4-months, and 8-months

CONTACTS AND LOCATIONS:
Locations (1):
- Rodney P. Joseph, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Metzendorf MI, Wieland LS, Richter B. Mobile health (m-health) smartphone interventions for adolescents and adults with overweight or obesity. Cochrane Database Syst Rev. 2024 Feb 20;2(2):CD013591. doi: 10.1002/14651858.CD013591.pub2. PMID 38375882
- [Derived] Joseph RP, Ainsworth BE, Vega-Lopez S, Adams MA, Todd M, Gaesser GA, Keller C. Cardiometabolic Risk Factors Among Insufficiently Active African American Women With Obesity: Baseline Findings From Smart Walk. J Cardiovasc Nurs. 2023 Mar-Apr 01;38(2):198-204. doi: 10.1097/JCN.0000000000000930. Epub 2022 Jul 5. PMID 35794781
- [Derived] Joseph RP, Ainsworth BE, Mathis L, Hooker SP, Keller C. Incorporating religion and spirituality into the design of community-based physical activity programs for African American women: a qualitative inquiry. BMC Res Notes. 2017 Oct 23;10(1):506. doi: 10.1186/s13104-017-2830-3. PMID 29058603